CLINICAL TRIAL: NCT00412503
Title: Phase 1 Study of Temozolomide Associated With Topotecan in Refractory or Relapsed Malignant Tumors in Children and Adolescents
Brief Title: Temozolomide in Association With Topotecan in Refractory or Relapsed Malignant Tumors in Children and Adolescents
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSET 1197
Record Dates: First submitted 2006-12-15; First posted 2006-12-18 (Estimated); Last update posted 2009-08-07 (Estimated); Status verified 2009-08

CONDITIONS: Refractory Tumors; Malignant Tumors
MeSH Terms: conditions — Neoplasms | interventions — Topotecan; Temozolomide

INTERVENTIONS:
Drug: Topotecan, Temozolomide

SUMMARY:
Long term survival can now be achieved in 75% of cases of pediatric cancers. However, some types of tumors (ie CNS tumors) or advanced stages (metastatic sarcomas/neuroblastomas) cannot be cured by any treatment. Thus, evaluation of new drugs or combinations are strongly needed. The recommended doses have been defined in children for TMZ (200 mg/m2/d x 5 d) and TPT (1.5 mg/m2/d x 5 d). Some preclinical and clinical studies have shown activity of both drugs in some pediatric cancers. Nevertheless, the association of the two drugs has never been evaluated. The study aims to determine Maximum Tolerated Dose and dose limiting toxicities of each drug when associated and to assess efficacy of the combination.

ELIGIBILITY:
Inclusion Criteria:

* histologically documented malignant tumor
* refractory or relapsing after conventional treatments and for which there is no curative treatment available
* life expectancy > 8 weeks
* no significant co-morbidity (NCI-CTC < 2)
* No organ toxicity
* no chemotherapy within the 4 previous weeks, 6 weeks for nitrosurea or radiotherapy

Exclusion Criteria:

* Hypersensibility to Topotecan and/or Temozolomide or to one of their compounds
* Hypersensibility to Dacarbazine (DTIC)
* Galactosaemia, Glucose and galactose malabsorption syndrom, deficiency in lactase

Ages: 6 Months to 21 Years | Sex: All
Age Groups: Child, Adult

PRIMARY OUTCOMES:
- To determine MTD and DLT of each drug

SECONDARY OUTCOMES:
To assess safety profile
To evaluate Pharmacokinetic of Temozolomide and Topotecan when associated
To assess the efficacy of the association

CONTACTS AND LOCATIONS:
Overall Officials: Herve Rubie, MD, Study Chair — University Hospital, Toulouse
Locations (1):
- Institut Gustave Roussy, Villejuif, Ille de France, France